CLINICAL TRIAL: NCT02492217
Title: Biomarkers Identification of Anti-TNF α Agent's Efficacy in Ankylosing Spondylitis Patients Using a Transcriptome Analysis and Mass Spectrometry
Brief Title: Biomarkers Identification of Anti-tumor Necrosis Factor (TNF) α Agent's Efficacy in Ankylosing Spondylitis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UniversidadeNL
Record Dates: First submitted 2015-07-03; First posted 2015-07-08 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; adalimumab; TNF-alpha agents; spondyloarthritis; biologic therapies; AS; biomarkers; efficacy prediction
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylarthritis | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adalimumab (Experimental): Adalimumab will be provided to trial participants as 0.8 ml single dose pre-filled syringes containing 40mg adalimumab each. A kit will be dispensed to he subject every two weeks, each kit containing one syringe.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab

SUMMARY:
To identify new candidate genes and proteins that are differentially expressed in responders' vs non-responders to anti-TNF alpha therapy at the several time points the investigators will use the transcriptomic and proteomic analyses. Demonstrate a link between gene expression and protein markers regarding prediction to anti-TNF alpha therapy efficacy.

ELIGIBILITY:
Inclusion Criteria:

* AS according to Portuguese Society of Rheumatology (SPR) guidelines (1984 modified New York Criteria, but allowing the use of MRI as imagiological criteria)
* Patient enrolment followed national guidelines for TNF antagonist use for the treatment of AS
* Adults between 18 to 75 years
* Ability to provide informed consent
* Corticosteroid therapy allowed (equivalent to ≤ 10 mg prednisone) and / or NSAID(nonsteroidal antiinflammatory drug), stable dose in 4 weeks before study initiation
* Adequate contraception (barrier or hormonal) in men and women of childbearing age (patients and their partners
* Adequate renal and hepatic function (2 times ULN)

Exclusion Criteria:

* Current pregnancy or breastfeeding
* Previous treatment with biologic DMARD's (disease-modifying antirheumatic drug)
* Intraarticular injections or infiltrations of extraaxial joints and tendons within 28 days before or at screening, or intraarticular injections of sacroiliac joints ≤ 28 days before screening
* History of rheumatic disorder other than AS
* Other forms of spondylarthritis than AS
* Any uncontrolled medical condition (e.g., uncontrolled diabetes mellitus, unstable ischemic heart disease)
* History or signs of demyelinating disease
* Malignancy (except for completely treated squamous or basal cell carcinoma)
* Moderate to severe heart failure (NYHA class III/IV) Positive serology for hepatitis B, hepatitis C, or human immunodeficiency virus
* Active or latent tuberculosis (TB) or histoplasmosis or other severe infections such as sepsis, and opportunistic infections
* Infections requiring hospitalization or intravenous treatment with antibiotics within 30 days or oral treatment with antibiotics within 14 days before enrollment
* Ankylosis of the spine (syndesmophytes presence at all levels from D12 to S1 in X-ray (XR) lateral view)
* Hypersensitivity to the active substance or to any of the excipients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Clinical response biomarkers (Assessment of Spondyloarthritis International Society (ASAS) 20 and Ankylosing Spondylitis Disease Activity Score (ASDAS) | 14 weeks
  To identify anti-TNF alpha clinical response biomarkers by microarrays and proteomics technology.

SECONDARY OUTCOMES:
QoL evaluation | 14 weeks
  To evaluate quality of life using ASQOL and SF-36 questionnaires
MRI progression | 14 weeks
  Rachis evaluation according to acute and structural lesions

CONTACTS AND LOCATIONS:
Overall Officials: Fernando M. Pimentel-Santos, MD, PhD, Study Chair — NOVA Medical School/Faculdade de Ciências Médicas; Jaime C. Branco, MD, PhD, Principal Investigator — NOVA Medical School/Faculdade de Ciências Médicas
Locations (1):
- Faculdade de Ciências Médicas da Universidade Nova de Lisboa, Lisbon, Portugal